CLINICAL TRIAL: NCT04002427
Title: A Phase I, Open-Label Study to Assess Mass Balance Recovery, Pharmacokinetics, Metabolite Profile & Metabolite Identification After Intravenous Microdose Administration of [14C]AZD7594 & Inhaled Administration of AZD7594 in Healthy Subjects
Brief Title: Mass Balance Recovery, Pharmacokinetics and Metabolite Profile and Identification of [14C]AZD7594
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3741C00010
Record Dates: First submitted 2019-04-18; First posted 2019-06-28 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only one study arm (Experimental): [14C]AZD7594 Solution for Infusion 5 µg/mL (1.1 kBq/mL)
  AZD7594 Inhalation Powder, SD3FL Inhaler
  Interventions: Drug: Intravenous Infusion; Drug: Inhaled dose

INTERVENTIONS:
Drug: Intravenous Infusion — 30 µg [14C]AZD7594 containing 6.7 kBq (180 nCi) carbon-14 (14C) as a 1 hour infusion.
Drug: Inhaled dose — A single inhalation on one occasion.

SUMMARY:
AZD7594 is in clinical development for the treatment of asthma.

This is a single centre, open-label, single period study in 6 healthy subjects, to determine the mass balance recovery and generate samples to enable metabolite profiling and structural identification of AZD7594.

Each subject will receive a single inhaled 792 µg nominal dose (720 µg delivered dose) of AZD7594 followed by an IV dose of 30 µg [14C]AZD7594 containing not more than (NMT) 6.7 kBq (180 nCi) carbon-14 (14C) as a 1 h infusion. The IV dose will be administered approximately 10 min after the inhaled dose. Subjects will remain resident in the clinical unit up to 168 h post dose (up to Day 8).

DETAILED DESCRIPTION:
This is a single centre, open-label, single period study in 6 healthy male and non-pregnant, non-lactating female subjects to determine the mass balance recovery after a single intravenous (IV) dose of [14C]AZD7594 and to generate samples to enable metabolite profiling and structural identification of AZD7594 in plasma, urine and faeces. It is planned to enrol 6 subjects to ensure data in at least 4 evaluable subjects. A subject will be considered evaluable if they have provided mass balance and PK samples for up to 48 h after drug administration.

Subjects will be screened for eligibility to participate in the study up to 28 days before dosing. Eligible subjects will be admitted to the clinical unit in the afternoon on the day before dosing (Day 1). Subjects will be dosed on the morning of Day 1 in the fasted state (8 h overnight fast). Before oral inhalation of AZD7594 using the Dry Powder Inhaler (DPI), all subjects must demonstrate their ability to use the DPI as intended. Subjects will receive training with an empty DPI at screening, Day -1 and pre-dose (optional) in accordance with study specific instructions. Each subject will receive a single inhaled 792 µg nominal dose (720 µg delivered dose) of AZD7594 followed by an IV dose of 30 µg [14C]AZD7594 containing 6.7 kBq (180 nCi) carbon-14 (14C) as a 1 h infusion. The infusion of the IV dose will be started approximately 15 min after the inhaled dose. Subjects will remain resident in the clinical unit up to 168 h post dose (up to Day 8).

Whole blood, plasma, urine and faeces will be collected from pre-dose until discharge (168 h post-dose; Day 8). Any accidental sources of elimination (eg emesis) will be collected and sent to the mass balance laboratory for total radioactivity analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male or non-pregnant, non-lactating female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venepuncture.
3. Have a body mass index of 18.5 to 35.0 kg/m2, and weigh at least 50 kg and no more than 100 kg, as measured at screening.
4. Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day).
5. Must be willing and able to communicate and participate in the whole study.
6. Must agree to adhere to the contraception requirements defined in Section 9.4 of the protocol.
7. Must demonstrate the ability to use the study inhalation device properly.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results of the volunteer's ability to participate in the study.
2. History or presence of clinically significant gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Subjects with Gilbert's syndrome or subjects with a history of cholecystectomy or gall stones.
5. Subjects with pregnant partners
6. Any confirmed clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the investigator.
7. Any confirmed clinically significant abnormal findings in vital signs or 12-lead ECG as judged by the investigator.
8. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
9. Has received any other new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose. Note: subjects consented and screened, but not randomised in this study or a previous Phase I study are not excluded.
10. Plasma donation within 1 month of screening or any blood donation/loss of more than 500 mL of blood during the 3 months prior to screening.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7594 or the formulation excipients including lactose. Hay fever is allowed unless it is active.
12. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission.
13. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
14. Females of childbearing potential who are pregnant or lactating (all female subjects must have a negative urine pregnancy test and screening and admission). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle stimulating hormone [FSH] concentration ≥40 IU/L).
15. Confirmed positive screen for drugs of abuse at screening or admission to the clinical unit or positive screen for alcohol at screening or admission to the clinical unit.
16. Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Subjects should stop using these herbal medications 14 days prior to administration of AZD7594.
17. Use of any prescribed or nonprescribed medication including antacids, H2 antagonists, PPI, analgesics (other than paracetamol/acetaminophen up to 4 g/day), vitamins and minerals during the 14 days prior to administration of AZD7594 or longer if the medication has a longer half-life (see Section 11.4 of the protocol). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
18. Known or suspected history of alcohol or drug abuse within the past 2 years or regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
19. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
20. Subjects who have previously been enrolled in this study.
21. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
22. Subjects who have been enrolled in an ADME study in the last 12 months
23. Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (ie during the screening period) minor medical complaints that may interfere with the interpretation of the study data or are considered unlikely to comply with the study procedures, restrictions and requirements.
24. History of infantile bronchiolitis, a history of asthma, adverse reaction or allergy to the inhaled medication or any excipients
25. Upper respiratory tract infection (excluding otitis media) within 14 days of the first study day, or lower respiratory tract infection within the last 3 months
26. Subjects who are unable to demonstrate their ability to fulfil the physical demands of the study
27. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
AZD7594 excreted (Ae) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of total radioactivity by measuring AZD7594 excreted (Ae)
AZD7594 excreted and expressed as a percentage of the administered dose (Fe) | Urine and faecal samples colected from pre-dose until 168 hours post-dose
  Assessment of total radioactivity by measuring AZD7594 excreted and expressed as a percentage of the administered dose (Fe)
Cumulative amount of AZD7594 excreted (CumAe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of total radioactivity by measuring the cumulative amount of AZD7594 excreted (CumAe)
Cumulative amount of AZD7594 excreted and expressed as a percentage of the administered dose (CumFe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of total radioactivity by measuring AZD7594 excreted and expressed as a percentage of the administered dose (CumFe)
Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of metabolites and structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of faecal samples from pre-dose until 168 hours post-dose
  Assessment of metabolites and structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of urine samples from pre-dose until 168 hours post-dose
  Assessment of metabolites and structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry

SECONDARY OUTCOMES:
Determination of routes and rates of elimination of [14C]AZD7594 | Collection of urine and faecal samples from pre-dose until 168 hours post-dose
  Assessment of total radioactivity by measuring AZD7594 excreted (Ae), cumulative recovery (Cumae), Ae as a percentage of the administered dose (Fe) and cumulative recovery expressed as a percentage of the dose (CumFe)
Determination of the chemical structure of the "major" metabolites of [14C]AZD7594 | Collection of urine adn faeces samples from pre-dose until 168 hours post-dose
  Structural identification by assessing liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Evaluation of whole blood:plasma concentration ratios for total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Assessment of total radioactivity by measuring AZD7594 in blood and plasma
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Time from dosing at which Cmax was apparent (tmax)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  The maximum observed plasma concentration (Cmax)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  The area under the concentration-time curve from dosing to the last measurable concentration (AUClast)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  The area under the concentration-time curve from dosing extrapolated to infinity (AUC0-inf)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  The percentage of AUC extrapolated beyond the last measured time point (AUC%extr)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  The terminal elimination rate constant calculated from the slope of the apparent elimination phase (λz)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  The apparent terminal elimination half-life (t½)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Total clearance (CL)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Volume of distribution (Vz)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Volume of distribution at steady state (Vss)
Assessment of the IV PK of [14C]AZD7594 and total radioactivity | Collection of plasma samples from pre-dose until 168 hours post-dose
  Mean residence time (MRT)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The time from dosing at which Cmax was apparent (tmax)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The maximum observed plasma concentration (Cmax)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The area under the concentration-time curve from dosing to the last measurable concentration (AUClast)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The area under the concentration-time curve from dosing extrapolated to infinity (AUC0-inf)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The percentage of AUC extrapolated beyond the last measured time point(AUC%exre)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The terminal elimination rate constant calculated from the slope of the apparent elimination phase (λz)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  The apparent terminal elimination half-life (t½)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  Apparent total clearance (CL/F)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  Apparent volume of distribution (Vz/F)
Assessment of the inhaled PK of AZD7594 | Collection of plasma samples from pre-dose until 168 hours post-dose
  Absolute bioavailability (F)
Number of adverse events (AE) | AEs recorded from the time of informed consent until discharge from the study (168 hours post-dose)
  Safety and tolerability assessed through incidence of AE

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences Limited (indemnified by
Locations (1):
- Research Site, Ruddington, United Kingdom